CLINICAL TRIAL: NCT05745870
Title: Effects of Creatine Supplementation and Resistance Training on Lean Mass, Sleep, Muscular Strength, and Perceived Menstrual Cycle Symptoms in Premenopausal Females
Brief Title: Creatine Supplementation and Resistance Training in Premenopausal Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Idaho (Other)
Responsible Party: Principal Investigator, Ann Brown, Associate Professor, University of Idaho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-170
Record Dates: First submitted 2023-02-06; First posted 2023-02-27 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Health Behavior
Keywords: Creatine monohydrate; resistance training; menstrual cycle; female physiology; body composition
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Creatine Monohydrate Supplementation (Experimental): Participants will consume 5g/d creatine monohydrate + 5g/d maltodextrin for 42 consecutive days
  Interventions: Dietary Supplement: Creatine Monohydrate Supplementation
- Placebo Supplementation (Placebo Comparator): Participants will consume 10g/d maltodextrin for 42 consecutive days
  Interventions: Dietary Supplement: Creatine Monohydrate Supplementation

INTERVENTIONS:
Dietary Supplement: Creatine Monohydrate Supplementation — Participants will consume 5g/d creatine monohydrate + 5g/d maltodextrin for 42 consecutive days

SUMMARY:
The goal of this clinical trial is to determine the effects of creatine monohydrate and resistance training on lean mass, sleep, muscular strength, and perceived menstrual cycle symptoms in untrained premenopausal females. The main questions it aims to answer are: 1) Does creatine monohydrate supplementation improve body composition, muscular strength, and sleep? 2) Does creatine monohydrate decrease perceived menstrual cycle symptoms compared to a placebo control?

Participants will be asked to consume creatine monohydrate daily for 42 consecutive days and well as perform a daily ovulation test. Pre and post testing will include assessments of urine specific gravity to determine hydration status, body composition testing, muscular strength testing and questionnaires.

Researchers will compare creatine monohydrate supplementation to a maltodextrin control to see if body composition, sleep, muscular strength, and perceived menstrual cycle symptoms are improved following 6-weeks.

DETAILED DESCRIPTION:
This study will be a 6 week creatine monohydrate and resistance training intervention with performance familiarization and pre and post testing. Participants will report to the Human Performance Laboratory (HPL), having fasted from alcohol, caffeine, and exercise for a minimum of 12-hours, for pre testing and to sign an informed consent explaining the procedures and potential risks and benefits of participation. Participants will then provide one urine sample to determine proper hydration status for body composition assessment. Next, participants will complete a physical activity readiness questionnaire (PARQ+) prior to performing any physical tasks. Participants will complete a daily menstrual cycle log, fatigue questionnaire, and health history survey. Prior to body composition testing, participants will complete a dual-energy x-ray apsorptiometry (DXA) scan consent for to ensure absence of pregnancy. Then, a full-body DXA scan will be completed along with an InBody bioelectrical impedance analysis. Following body composition testing, participants will be fitted for an Oura ring to track their sleep. Lastly, muscular strength will be assessed using the Tonal. Following a 5-minute full-body warm up, 1-repetition maximum will be determined using two upper body and two lower body exercises at maximal effort. Upon conclusion of pre-testing, participants will be randomized into two groups: 1) creatine monohydrate (5g/d creatine monohydrate + 5g/d maltodextrin) or 2) placebo (10 g/d maltodextrin) for 42 consecutive days. Participants will visit the HPL daily to consume their respective supplement as well as provide a urine sample for ovulation status determination. Additionally, participants will complete two resistance training sessions on non-consecutive days using the Tonal per week for 6-weeks. Following 6-weeks, post-testing will occur and includes the same procedures as pre-testing.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal females 18-25 yrs
* able to resistance train with no contraindications to exercise testing

Exclusion Criteria:

* premenopausal female taking hormonal contraceptives
* premenopausal females who are resistance training >2x/wk
* premenopausal females who consume creatine monohydrate

Ages: 18 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Premenopausal female not taking contraceptives
Enrollment: 27 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Body Composition | 42 days
  Change in lean mass (kg, %) using a DXA scan from baseline after 42 days
Sleep | 42 days
  Change in sleep (hours, minutes, REM) using the Oura Ring application tracking from baseline after 42 days
Muscular Strength | 42 days
  Change in muscular strength (1-repetition maximum) using the Tonal from baseline after 42 days
Perceived Menstrual Cycle Symptoms | 42 days
  Change in perceived menstrual cycle symptoms (fatigue, cramping, bloating) using menstrual cycle questionnaires from baseline after 42 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Idaho, Moscow, Idaho, United States

IPD SHARING:
Plan to Share IPD: No